CLINICAL TRIAL: NCT04494802
Title: The Influence of LMA Cuff Pressure on Oropharyngeal Leak Pressure and Gastric Insufflation Assessed by Ultrasound in Pediatric Patients
Brief Title: The Influence of LMA Cuff Pressure on Gastric Insufflation Assessed by Ultrasound in Pediatric Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gastric insufflation
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Aspiration
MeSH Terms: interventions — Lower Body Negative Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- higher pressure (Placebo Comparator): During the operation, cuff pressure of LMA flexible is maintained to 50cmH2O
  Interventions: Behavioral: higher pressure
- lower pressure (Experimental): During the operation, cuff pressure of LMA flexible is maintained to 30cmH2O
  Interventions: Behavioral: lower pressure

INTERVENTIONS:
Behavioral: lower pressure — During the operation, cuff pressure of LMA flexible is maintained to 30cmH2O
  Arms: lower pressure
Behavioral: higher pressure — During the operation, cuff pressure of LMA flexible is maintained to 50cmH2O
  Arms: higher pressure

SUMMARY:
Cuff inflation up to the maximum cuff pressure when using LMA flexible can cause sore throat and discomfort after the surgery, and if the surgery is unexpectedly prolonged, there can be a side effect that can cause ischemic damage around the neck. If keeping cuff pressure low will not increase gastric insufflation and there is no change in other outcome variables, keeping it low may have a positive effect on anesthesia management and outcome in children.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia with LMA flexible

Exclusion Criteria:

* Unstable vital sign, significant arrhythmia or hypotension, Shock
* anticipated difficult intubation or the patient who have facial deformity
* high risk of aspiration
* recent upper respiratory tract infection history

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastric insufflation(antrum) | During the surgery(up to 3 hours)
  Incidence of gastric insufflation which was recognized in gastric antrum with ultrasound

SECONDARY OUTCOMES:
The size of gastric antrum and body | During the surgery(up to 3 hours)
  The size of gastric antrum and body assessed immediately after insertion of LMA flexible and after finishing the surgery
Time for insertion of LMA flexible | During the anesthesia induction(up to 1 hour)
  Time for insertion of LMA flexible
Success rate of insertion of LMA flexible | During the anesthesia induction(up to 1 hour)
  Success rate of insertion of LMA flexible
The number of insertion attempt | During the anesthesia induction(up to 1 hour)
  The number of insertion attempt
The number and the type of additional manipulation for successful ventilation | During the surgery(up to 3 hours)
  The number and the type of additional manipulation for successful ventilation
Ease of insertion of LMA flexible | During the anesthesia induction(up to 1 hour)
  Ease of insertion of LMA flexible(very easy, easy, moerate, difficult, very difficult)
Incidence of gastric insufflation(body) | During the surgery(up to 3 hours)
  Incidence of gastric insufflation which was recognized in gastric body with ultrasound
Incidence of gastric insufflation recognized with the ausculation | During the surgery(up to 3 hours)
  Incidence of gastric insufflation recognized with the ausculation after finishing surgery
peak pressure observed before, during, after surgery | During the surgery(up to 3 hours)
  peak pressure observed before, during, after surgery
oropharyngeal leak pressure | During the surgery(up to 3 hours)
  oropharyngeal leak pressure will be assessed by setting the APL valve of the circle system at 30 cmH2O with fresh gas flow of 3 L/min after the surgery
the complication rate | During the surgery and after surgery (up to 6 hours)
  the complication rate such as desaturation, blood staining of LMA flexible, hoarseness, dental/lip/tongue injury, aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided